CLINICAL TRIAL: NCT06445426
Title: Cystometry Using a Novel Microsensor System in Patients With Neurogenic Bladder Dysfunction
Acronym: PEPRE2
Status: Completed | Type: Observational
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: SINTEF MiNaLab (Unknown); University of Oslo (Other)
Responsible Party: Principal Investigator, Thomas Glott, Medical director, Sunnaas Rehabilitation Hospital
Other Study IDs: SUPRE
Record Dates: First submitted 2022-08-05; First posted 2024-06-06 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Spinal Cord Injuries; Urinary Bladder, Neurogenic
Keywords: Urodynamics
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Simulataneous bladder pressure recording: In all patients recruited, the pressure will be recorded simultaneously with the conventional and novel pressure recording systems in the bladder. The procedure will be done according to the International Continence Society's (ICS) recommended indications for the procedure.
  Interventions: Device: Cystometry

INTERVENTIONS:
Device: Cystometry — The procedure will be done according to the International Continence Society's (ICS) recommended indications for the procedure. The investigational device is inserted into a 12F single-use hydrophilic catheter. After correct positioning is verified by ultrasound and x-ray, the investigational device is released from the insertion catheter. The insertion catheter is then carefully removed, securing the correct positioning of the investigational device inside the bladder. The investigational device is connected to a data logger. In the conventional device, the intravesical pressure is recorded using a water perfused 3F catheter with a 3 ml/hour perfusion rate. The 3F catheter is hooked on an 8F catheter to facilitate introduction into the bladder. The catheters used for pressure transmission are connected to external transducers and a computer with software processing the recording
  Other Names: Pressure measurement in the urinary bladder

SUMMARY:
The aim of this study is to assess the feasibility and safety of a novel system for percutaneous measurement of bladder pressure. This system enables minimally invasive procedures and high-quality recordings, offering a sampling rate and synchronization surpassing traditional methods. The pressure sensor system has the potential to be developed into a low-cost method suitable for mass production. The study will include a sample of convenience of up to 40 subjects. Pressure will be recorded simultaneously in the bladder using both the conventional and novel pressure recording systems. This simultaneous recording method will provide a direct comparison of pressure recordings between the two systems. Subjects will be examined for any subjective or objective adverse events.

DETAILED DESCRIPTION:
The aim of this study is to assess the feasibility and safety of a novel system for measurement of bladder pressure. The system facilitates a minimally invasive procedure, enabling high-quality recordings with a sampling rate and synchronization that surpass conventional standards. The pressure sensor system has potential to be developed into a low-cost method with mass production. In patients with spinal cord injury and neurogenic bladder dysfunction, measurement of pressure in the bladder (cystometry) is mandatory to evaluate risk factors and assess treatment options. This novel system consists of a micro electro mechanical system (MEMS) integrated in a hollow flexible tube made out of biocompatible material. Recording from this sensor catheter is transmitted to specialized electronic and digital devices for processing. Due to a sensor catheter with a diameter less than 1.0 mm, it is possible to perform transurethral cystometry using a simple minimally invasive technique. The study goal is to compare the simultaneous measurement of the conventional water perfused system compared to a novel pressure sensor system during cystometry. produce high-quality recordings with a higher than conventional sampling rate. The study will include a sample of convenience of up to 40 subjects. The pressure will be recorded simultaneously with the conventional and novel pressure recording system in the urinary bladder. The simultaneous recording with the novel and the conventional method will provide a direct comparison of simultaneous recording of pressure between the two systems. Patients will be examined for subjective or objective adverse events. The sample size is too small for comparison of validity of the two methods in clinical practice. However, the study should be able to conclude on reliability. Thus, pressure measurements will be assessed with both methods during cystometry in up to 40 subjects. Given the technical specifications, the measurements are expected to be nearly identical, thereby ensuring reliability. The study is not intended to provide conclusive results on the comparison between conventional water perfused recording and the novel MEMS pressure system. However, results from this initial study will be the basis for further studies with sufficient power to validate conventional versus novel MEMS technique.

ELIGIBILITY:
Inclusion Criteria:

* Documented traumatic or non-traumatic spinal cord injury
* Documented neurogenic bladder dysfunction by previous cystometry
* More than 3 months after injury
* Subject is able to communicate in Norwegian
* Subject is able and willing to sign informed consent
* Subject is able to complete all study requirements

Exclusion Criteria:

* History or evidence of previous urological or lower abdominal abnormalities from disease or surgery
* Use of anti-platelet or anti-coagulant other than low molecular weight heparin or acetylsalicylic acid which cannot be discontinued
* Symptomatic urinary tract infection
* Hemophilia or other clotting disorders that cause bleeding diathesis
* Any condition or situation, which, in the investigator's opinion, puts the subject at significant risk, could confound the study results, or may interfere significantly with the subject's participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from patients with chronic spinal cord injury (SCI) admitted for cystometry at Sunnaas Hospital´s urodynamic laboratory. All subjects will have a clinical indication for cystometry.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Bladder pressure | 24 hours
  The bladder pressure recorded simultaneously by a conventional clinical system and the prototype will be used for a systemstic comparison analysis in the time-amplitude and the time-frequency domains.

OTHER OUTCOMES:
Advert effects monitoring and resolution | 72 hours
  Subjects will be examined for any subjective or objective adverse events. The transurethral technique is well-known, and the complication rates are very low. However, there are known complications such as urinary tract infection, hematuria, pain, retention, and autonomic dysreflexia in tetraplegics. Subjects will be routinely examined for all these conditions, and if any of them occur, adequate treatment will be initiated according to hospital guidelines. The small-sized sensor tube (Ø ≈ 1.2 mm) provides a minimally invasive clinical procedure. In case of perforation, the lesion will be small.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnaas Rehabilitation Hospital, Oslo, Nesoddtangen, Norway

IPD SHARING:
Plan to Share IPD: No